CLINICAL TRIAL: NCT01067664
Title: The Effect of Serum Progesterone Levels on the Day of hCG Administration on the Probability of Pregnancy in Patients Treated by IVF Using GnRH Antagonists and Recombinant Gonadotrophins
Brief Title: Prognostic Value of Progesterone for In Vitro Fertilization (IVF) Outcome
Acronym: PROG2
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Basil C. Tarlatzis, MD, PhD, 1st Dept. of Obstetrics and Gynaecology, Medical School, Aristotle University of Thessaloniki
Other Study IDs: UHR-7
Record Dates: First submitted 2009-11-01; First posted 2010-02-11 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-06

CONDITIONS: Subfertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 6ml of serum will be frozen and stored for later analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing IVF with rFSH and GnRH antagonists

SUMMARY:
This observational study attempts to investigate the potential role of serum progesterone levels on the day of hCG administration (thus, the end of the follicular phase) on the probability of pregnancy, in patients undergoing IVF with the use of GnRH antagonists and recombinant gonadotrophins.

There has been evidence, that increased serum levels of progesterone are associated with a decreased probability of pregnancy after IVF.

This study will attempt to explore the role of progesterone on the outcome of IVF, by closely monitoring its levels during the late follicular phase.

ELIGIBILITY:
Inclusion Criteria:

* Age < 40 years
* Basal FSH < 12 IU/L
* Basal P < 1.6 ng/mL

Exclusion Criteria:

* Presence of cystic formations at the ovaries during the basal ultrasound scan (prior the initiation of stimulation)
* Women with polycystic ovaries syndrome (PCOS)
* Women with Stage III-IV Endometriosis
* Women with a pathological condition of the adrenal glands

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing ovarian stimulation with the use of rFSH and GnRH antagonists for in-vitro fertilization.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy, defined as ultrasound evidence of fetal heart activity at 6-8 weeks of gestation | At 6-8 weeks of gestation

SECONDARY OUTCOMES:
Pregnancy (defined as a b-hCG> 25 IU/L) | 12 days after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Basil C Tarlatzis, MD, PhD, Principal Investigator — 1st Dept. of Obstetrics and Gynaecology, Medical School, Aristotle University of Thessaloniki; Christos A Venetis, MD, MSc, Principal Investigator — Unit for Human Reproduction, 1st Dept. of Obstetrics and Gynaecology, Medical School, Aristotle University of Thessaloniki
Locations (1):
- Unit for Human Reproduction, 1st Dept. of Obstetrics and Gynaecology, Medical School, Aristotle University of Thessaloniki, Thessaloniki, Greece